CLINICAL TRIAL: NCT01618500
Title: Computerised Testing of Cognitive Response to Cerebrospinal Fluid Shunting in Idiopathic Normal Pressure Hydrocephalus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Anders Behrens, M.D., M.Sc., Umeå University
Other Study IDs: 2011-47-31M
Record Dates: First submitted 2012-06-11; First posted 2012-06-13 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Normal Pressure Hydrocephalus
Keywords: Normal Pressure Hydrocephalus; Neuropsychological Test; Assessment of cognitive disorders/dementia; Neuropsychological assessment
MeSH Terms: conditions — Hydrocephalus, Normal Pressure; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- INPH-patients: Inclusion criteria
  Older than 60 years of age "Probable INPH" according to the NIH guidelines Planned shunt surgery based on a diagnosis of INPH.
  Exclusion criteria
  Known cause for hydrocephalus (i.e., secondary NPH). Medical condition preventing cognitive testing (e.g. deafness, blindness).
  Patients not considered for shunt operation.

SUMMARY:
A novel computerised neuropsychological test battery for normal pressure hydrocephalus (NPH) has been developed. The aim is to provide the clinician with a free of charge, standardized tool, assessing the cognitive decline or improvements in the cognitive domains specific for NPH. Results from the battery indicate good reliability and validity for the computerized tests

Results from the computerised battery seems promising. However, ability for the battery to detect cognitive improvements after a shunt operation remains to be tested.

Study objectives

1. Improvement after shunt. The aim of this study is to evaluate the effects of shunting on neuropsychological performance in NPH patients, using a computerized battery.
2. Feasibility. The ability to complete the test battery by the intended patient group will be tested.
3. Baseline profile. Baseline scores for NPH-patients will be compared to scores of healthy individuals (from previous study).

ELIGIBILITY:
Inclusion Criteria:

* Older than 60 years of age

"Probable INPH" according to the NIH guidelines

Planned shunt surgery based on a diagnosis of INPH.

Exclusion Criteria:

* Known cause for hydrocephalus (i.e., secondary NPH). Medical condition preventing cognitive testing (e.g. deafness, blindness).

Patients not considered for shunt operation.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eighty INPH-patients. Consecutively included.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Neuropsychological outcome | 4.5 ± 1.5 months
  INPH patients, who are shunt candidates, will complete a computerized battery at two occasions: (1) hospital admission (Baseline) at most 1 month prior to surgery, and (2) 4.5 ± 1.5 months after shunt operation (Post-Shunt).

SECONDARY OUTCOMES:
Mini mental state Examination | 4.5 ± 1.5 months
  INPH patients, who are shunt candidates, at each center will complete the Mini Mental State Examination at: (1) hospital admission (Baseline) at most 1 month prior to surgery, and (2) 4.5 ± 1.5 months after shunt operation (Post-Shunt).
Feasibility | 4.5 ± 1.5 months
  The number of patients who are able to complete individual subtests and the entire battery, will be monitored.
Baseline cognitive profile compared to healthy
  The baseline cognitive profile of INPH-patients will be compared to healthy individuals (from previous study).

CONTACTS AND LOCATIONS:
Locations (4):
- Ålborg University Hospital, Aalborg, Denmark
- Sweden (3):
  - Linköping University Hospital, Linköping
  - Umeå University, Umeå
  - Akademiska sjukhuset, Uppsala

REFERENCES:
- [Derived] Behrens A, Elgh E, Leijon G, Kristensen B, Eklund A, Malm J. The Computerized General Neuropsychological INPH Test revealed improvement in idiopathic normal pressure hydrocephalus after shunt surgery. J Neurosurg. 2019 Feb 8;132(3):733-740. doi: 10.3171/2018.10.JNS18701. Print 2020 Mar 1. PMID 30738407